CLINICAL TRIAL: NCT06475430
Title: Evaluation of the Effectiveness of Fecal Microbiota Transplantation in the Treatment of Patients With Severe Low Anterior Resection Syndrome (LARS)
Brief Title: Fecal Microbiota Transplantation in the Treatment of Major LARS
Acronym: FMT-LARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Fan Liu, Fan Liu, Peking University People's Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BaS-2406
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Low Anterior Resection Syndrome; Fecal Microbiota Transplantation
Keywords: low anterior resection syndrome; bowel function; fecal microbiota transplantation; intestinal microbiota
MeSH Terms: conditions — Low Anterior Resection Syndrome | interventions — Fecal Microbiota Transplantation; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal flora transplantation group (Experimental)
  Interventions: Biological: fecal microbiota transplantation
- Formulated probiotics group (Active Comparator)
  Interventions: Dietary Supplement: Formulated probiotic supplements

INTERVENTIONS:
Biological: fecal microbiota transplantation — During the treatment, a colonoscopic colonic catheter will be placed via the anus, with the experimental group receiving FMT solution matched to the patient's microbiota for intra-intestinal administration.
  Other Names: FMT
  Arms: Fecal flora transplantation group
Dietary Supplement: Formulated probiotic supplements — During the treatment, a colonoscopic colonic catheter will be placed via the anus, with the control group receiving a standardized probiotic formula.
  Other Names: probiotic
  Arms: Formulated probiotics group

SUMMARY:
Randomized trial to assess FMT efficacy in improving bowel function for major LARS patients. 40 subjects, blinded, randomized to FMT or probiotics. Pre-post 16S sequencing, 4-week follow-up for bowel symptoms, 8-week microbiota analysis.

DETAILED DESCRIPTION:
This study is a rigorous single-center, prospective, double-blinded, randomized controlled trial, aiming to evaluate the effectiveness of fecal microbiota transplantation (FMT) in improving bowel function for patients with major low anterior resection syndrome (LARS). A total of 40 subjects are planned to be recruited and randomly assigned to the experimental group and the control group at a 1:1 ratio. Prior to treatment, all subjects will undergo 16S sequencing of intestinal microbiota to assess their intestinal microecological status. During the treatment, a colonoscopic colonic catheter will be placed via the anus, with the experimental group receiving FMT solution matched to the patient's microbiota for intra-intestinal administration, while the control group will receive a standardized probiotic formula. To ensure the impartiality of the study, both patients and researchers administering the medication will be blinded to the trial drugs. The study will continuously observe and record bowel symptoms after 4 weeks of treatment as well as 16S sequencing results of intestinal microbiota after 8 weeks. Upon the completion of the entire study, the blinding will be revealed, and the results will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years old, regardless of gender; Patients with rectal cancer who have undergone total mesorectal excision (TME) and sphincter-preserving surgery, and the postoperative period is more than 3 months; Patients with a LARS score of 21 to 42; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1; Expected survival period ≥ 1 year; Voluntarily sign a written informed consent form.

Exclusion Criteria:

- Patients with pre-operative symptoms of fecal and urinary incontinence; Patients who have undergone pelvic surgery or LAR due to non-cancerous reasons; Patients who have undergone pelvic radiotherapy; Patients with prophylactic ostomy; Patients who have used any antibiotic medication, probiotic products, or prebiotic products in the past 4 weeks; Patients who have regularly used laxatives in the past two weeks; Pregnant or lactating women; Human immunodeficiency virus (HIV) positive; Known history of active pulmonary tuberculosis (TB). Subjects suspected of having active TB require chest X-ray, sputum examination, and exclusion based on clinical symptoms and signs; Untreated patients with chronic hepatitis B or HBV carriers with HBV DNA exceeding 500 IU/mL, or patients with active hepatitis C should be excluded. Non-active HBsAg carriers, treated and stable hepatitis B patients (HBV DNA < 500 IU/mL), and cured hepatitis C patients can be enrolled. For subjects with positive HCV antibodies, only those with negative HCV RNA test results are eligible to participate in the study; Known history of psychiatric drug abuse, alcoholism, and drug abuse; Patients with cognitive impairment; Any situation where the investigator believes the participant should be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
bowel function | 4 weeks and 8 weeks
  LARS score
Shannon index | 8 weeks
  biodiversity monitoring

IPD SHARING:
Plan to Share IPD: No